CLINICAL TRIAL: NCT05441007
Title: The Effect of Hypercapnia and Hypoxia on Physiological Parameters During Short-term Breathing Experiment
Brief Title: The Effect of Hypercapnia on Physiological Parameters During Short-term Breathing
Acronym: HYPERCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CTU HYPERCO
Record Dates: First submitted 2022-06-25; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Hypoxia; Hypercapnia; Cardiac Output, High
Keywords: Cardiac Output; Perfusion index; Pulse oximetry
MeSH Terms: conditions — Hypoxia; Hypercapnia; Cardiac Output, High

STUDY DESIGN:
Intervention Model Description: Interventional single blinded randomized crossover prospective study. All participants go through all study arms, in random order.
Who Masked: Participant
Masking Description: The participant undergoes all three phases of the experiment and the participant does not know which one is it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypoxic (Experimental): Participants inhale ambient air, the hypoxic gas mixture, and ambient air.
  Interventions: Other: Hypoxic
- Hypercapnic (Experimental): Participants inhale ambient air, the hypercapnic gas mixture, and ambient air.
  Interventions: Other: Hypercapnic
- Hypoxic and Hypercapnic (Experimental): Participants inhale ambient air, the hypoxic and hypercapnic gas mixture, and ambient air.
  Interventions: Other: Hypoxic and Hypercapnic

INTERVENTIONS:
Other: Hypoxic — Hypoxic gas mixture Gas mixture of 10% O2 and 90% N2 for six minutes.
  Arms: Hypoxic
Other: Hypercapnic — Hypercapnic gas mixture Gas mixture of 21% O2, 5% CO2 74% N2 for six minutes.
  Arms: Hypercapnic
Other: Hypoxic and Hypercapnic — Hypoxic and Hypercapnic gas mixture Gas mixture of 10% O2, 5% CO2 85% N2 for six minutes.
  Arms: Hypoxic and Hypercapnic

SUMMARY:
The aim of the project is to evaluate the effect of hypercapnia on physiological parameters in a healthy person during short-term hypoxia and hypercapnia.

DETAILED DESCRIPTION:
Hypercapnia causes changes in physiological parameters at various levels throughout the body. The study aims to evaluate the effect of hypercapnia on physiological parameters in a healthy person during short-term hypoxia and hypercapnia. It is an intervention prospective study that will be conducted at the Faculty of Biomedical Engineering on healthy volunteers. All the volunteers undergo three different phases in random order. The individual phases differ in the breathed mixture of oxygen, nitrogen and carbon dioxide gases. Non-invasive measurements of physiological parameters, especially blood oxygen saturation, perfusion index and cardiac output, will be performed continuously during the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* injury to the upper limbs or hands that could affect the peripheral perfusion
* diabetes
* hypotension or hypertension

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Cardiac output due to the induced hypoxia and hypercapnia | 1 hour
  Based on the induced hypoxia, hypercapnia or combination of hypoxia and hypercapnia, Cardiac output will change
Changes in Perfusion index due to the induced hypoxia and hypercapnia | 1 hour
  Based on the induced hypoxia, hypercapnia or combination of hypoxia and hypercapnia, Perfusion index will change

CONTACTS AND LOCATIONS:
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No